CLINICAL TRIAL: NCT02315521
Title: Validation of the Standardized Prenatal Clinical Management of Fetuses With Lower Urinary Tract Obstruction (LUTO)
Brief Title: Standardized Prenatal Clinical Care for LUTO
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Michael A Belfort, Professor and Chairman, Department of Obstetrics and Gynecology, Baylor College of Medicine
Other Study IDs: BCM H-35770
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Urethral Obstruction
Keywords: lower urinary tract obstruction; posterior urethral valves; urethral atresia; Prune Belly Syndrome; Megalo-urethra; Fetal renal function; Prenatal Diagnosis; Ultrasound
MeSH Terms: conditions — Urethral Obstruction; Prune Belly Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: Fetuses with LUTO before 18 weeks
  Interventions: Procedure: Fetal Intervention for LUTO
- Group 2: Fetuses with LUTO between 18 and 30 weeks
  Interventions: Procedure: Fetal Intervention for LUTO
- Group 3: Fetuses with LUTO between 30 and 34 weeks
  Interventions: Procedure: Fetal Intervention for LUTO
- Group 4: Fetuses with LUTO after 34 weeks

INTERVENTIONS:
Procedure: Fetal Intervention for LUTO — Fetal vesico-amniotic shunting placement consists in placing a shunt (stent) percutaneously from fetal bladder to the amniotic cavity under ultrasound guidance.
  Fetal cystoscopy will be performed using a thin scope that will be introduced to the fetal bladder for evaluation of the cause of the obstruction and ablation of the posterior urethral valves.
  Other Names: Fetal vesico-amniotic shunting; Fetal cystoscopy
  Groups: Group 1; Group 2; Group 3

SUMMARY:
The investigators propose a standardized prenatal management, based on the scientific evidence published in the literature, to manage prenatally fetuses with lower urinary tract obstruction (LUTO). The present study is a prospective registry that will evaluate and validate this standardized prenatal management for LUTO.

DETAILED DESCRIPTION:
Patients with LUTO will come for clinical evaluation as part of the standard clinical care at the our Fetal Center. The standardized prenatal management of plan for fetuses with LUTO is described in details bellow.

All pregnant women carrying fetuses with LUTO are assigned to the nurse coordinator and the prenatal records are obtained. The multidisciplinary team (maternal-fetal intervention team, pediatric urologists, pediatric nephrologist, neonatologist, genetic counselors and fetal cardiologists) will be notified. A one-day visit is planned with the following: 1. a fetal comprehensive ultrasound is scheduled for the confirmation of the diagnosis, investigation of associated anomalies and evaluation of prognostic factors; 2. a genetic counseling is performed and fetal invasive tests (FISH/fetal karyotype/fetal CMA) are offered to the patients; 3. Fetal echocardiogram is also performed to evaluate the presence of associated cardiac anomalies and the fetal cardiac function; 4. A consultation with the Fetal Intervention team (maternal-fetal specialty) is scheduled as well. Additionally, maternal and fetal samples (maternal blood, amniotic fluid, fetal blood, and fetal urine) will be collected as part of the standardized clinical management. We plan to investigate the analysis of those samples, and to also collect more samples for banking to be used in future studies.

If the gestational age is less than 18 weeks and isolated LUTO is confirmed on ultrasonography, patient is giving the option for prenatal expectant management, or fetal intervention or termination of pregnancy. If patient elects to proceed with fetal intervention, vesico-amniotic shunting is performed and patient is followed by ultrasound once a week. In case the shunt migrates or seems to be obstructed, we will offer repeating the procedure to the patient. If patient elects to proceed with expectant management, follow-up will be every 4 weeks. Delivery date and type of delivery depend on the obstetrical indications.

For fetuses at gestational age greater than 18 and less than 30 weeks, if oligohydramnios is present, investigation of fetal renal biochemistry is offered. In case of favorable fetal renal biochemistry, vesico-amniotic shunt is offered as a fetal therapeutic intervention. In case the fetal urinary biochemistry is considered not favorable, then we will repeat the urinary examination in 24 hours. If the fetal urinary biochemistry is still not favorable, we will repeat the examination for the last time (maximum of 3 times). If it is still not favorable, then fetal vesico-amniotic shunt is not offered. However, if a fetal urinary examination reveals improvement favorable urinary biochemistry), fetal vesico-amniotic shunting is considered. Prenatal follow-up and delivery follow the same algorithm described previously.

If gestational age is greater than 30 weeks and less than 34 weeks and isolated LUTO is diagnosed, fetal intervention is offered if oligohydramnios is present. If no oligohydramnios is identified, no fetal intervention is offered and patient is followed until delivery. Delivery date and type of delivery depend on the obstetrical indications.

For those fetuses with gestational age greater than 34 weeks, if oligohydramnios is present, pre-term delivery is indicated. If a normal amount of amniotic fluid is seen, patient is followed weekly by ultrasound examination and delivery is at term.

Fetuses with other associated anomalies independent from the gestational age will undergo further investigation with fetal magnetic resonance imaging and evaluation by the multidisciplinary team.

All infants with LUTO will have the same routine standard clinical care. All infants with LUTO are evaluated postnatally by the pediatric urology and nephrology services and may need surgical intervention. At birth, the clinical evaluation will include a renal ultrasound, voiding cysto-urethrogram (VCUG) as well as clinical laboratory examinations such as serum creatinine, sodium, calcium, potassium and chloride, and a urine analysis will be performed as part of the standard clinical care. The infant will be followed every 6 months up until 24 months of life, and then annually afterwards. Information from these routine examinations will be collected and documented.

ELIGIBILITY:
Inclusion Criteria:

- Pregnant women whose fetuses have diagnosis of LUTO independently from the gestational age at diagnosis.

Exclusion Criteria:

* Presence of abnormal chromosomal/genetic disease
* Presence of other associated structural anomaly that is not part of LUTO.

Ages: 11 Weeks to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All pregnant women referred to our Fetal Center with confirmed diagnosis of fetal LUTO. The diagnosis of fetal LUTO is based on the presence of enlarged bladder and bilateral hydronephrosis.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Survival rate | Survival rate since prenatal period to 24 months of life
  The survival rate from the prenatal period up to 24 months of life will be evaluated

SECONDARY OUTCOMES:
Postnatal renal function at 6 months of life | During neonatal period and at 6 months of life
  Renal function during neonatal period and at 6 months of life will be evaluated by analyzing the serum creatinine, weight and height, renal function, bladder function, lung disease, need for dialysis and transplantation, arterial hypertension, incontinence and developmental delay
Postnatal renal function at 12 months of life | During neonatal period and at 12 months of life
  Renal function during neonatal period and at 12 months of life will be evaluated by analyzing the serum creatinine, weight and height, renal function, bladder function, lung disease, need for dialysis and transplantation, arterial hypertension, incontinence and developmental delay
Postnatal renal function at 24 months of life | During neonatal period and at 24 months of life
  Renal function during neonatal period and at 24 months of life will be evaluated by analyzing the serum creatinine, weight and height, renal function, bladder function, lung disease, need for dialysis and transplantation, arterial hypertension, incontinence and developmental delay

CONTACTS AND LOCATIONS:
Overall Officials: Michael Belfort, MD PHD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital - Pavilion for Women, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No